CLINICAL TRIAL: NCT00361933
Title: Clinical and Virologic Response to HHV-8 Associated Multicentric Castleman's Disease to Valganciclovir
Brief Title: Valganciclovir to Treat HHV-8 Associated Multicentric Castleman's Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Research never begun.
Sponsor: University of Washington (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Corey Casper, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30618; VAL096
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Giant Lymph Node Hyperplasia
MeSH Terms: conditions — Castleman Disease | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — valganciclovir open label, two 450mg tablets orally, twice a day
  Other Names: Valcyte

SUMMARY:
The purpose of the study is to learn whether people who are experiencing an MCD (multicentric Castleman's Disease) flare will improve after taking valganciclovir. MCD is a type of inflammatory disease associated with Human Herpesvirus 8 (HHV-8). Valganciclovir is FDA approved for treating a different type of Human Herpesvirus, but not approved for the treatment of HHV-8. It is therefore considered experimental in this study.

DETAILED DESCRIPTION:
All participants will undergo an initial screening appointment. At this visit, participants will be tested for Human Herpesvirus 8 (HHV-8), the virus that is associated with MCD, and we will review participants' medical history and medical records to determine whether he/she has MCD. If participants do not live within the Seattle area, this visit may occur over the phone.

Those who qualify for the study will be followed for up to 2 years. During that 2 year period, participants will be asked to collect oral swabs once a week and have blood drawn monthly. If subjects do not live within the Seattle-area, they will be asked to ship these samples to UW for testing. We will provide subjects with instructions for these shipments. This will be done at no cost to the participant.

If during the 2 year period the participant experiences a MCD flare, he/she will be admitted to the University of Washington Medical Center's Clinic Research Center for 14-days. If the participant does not live within the Seattle-area, all travel expenses will be covered.

The study will enroll a total of 8 patients who will receive open-label valganciclovir for 14-days. Everyday during the hospitalization, participants will have blood drawn (to check your HHV-8 levels), 1 oral swab will be collected and a general physical exam will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Negative pregnancy test (for female participants)
* Diagnosis of MCD for over one year, with a history of at least one MCD recurrence annually
* Evidence of infection with HHV-8
* A willingness to travel and reside temporarily in Seattle for completion of the study protocol.
* For HIV-infected participants, a stable antiretroviral regimen for the past 6 months

Exclusion Criteria:

* Concurrent Kaposi sarcoma or non-hodgkin's lymphoma
* A history or evidence of CMV disease
* Hypersensitivity to ganciclovir or valganciclovir
* Use of high-dose acyclovir (>800 mg bid), valacyclovir (>1000 mg qd) or famciclovir (>1000 mg qd), ganciclovir, foscarnet, or cidofovir
* Neutropenia (ANC <1500)
* Renal insufficiency with serum creatinine > 1.5 mg/ml or CrCl < 60
* AST or ALT > 5 times upper limit of normal
* Concurrent administration of medications which are often associated with severe neutropenia or thrombocytopenia (i.e., chemotherapy, etc)
* Concurrent administration of probenecid or didanosine.
* Inability to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Time to improvement | 14 days
One-log reduction in HHV-8 peripheral blood viral load | 14 days

SECONDARY OUTCOMES:
Safety and tolerability of valganciclovir | 14 days
Proportion of patients resolving symptoms by 4 days | 14 days
HHV-8 detection in the plasma or oropharynx | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Corey Casper, MD, MPH, Principal Investigator — University of Washington